CLINICAL TRIAL: NCT02455206
Title: Effect of Counseling During Pulmonary Rehabilitation on Self-determined Motivation Towards Physical Activity in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Counseling During Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich University of Applied Sciences (Other)
Collaborators: Kantonsspital Winterthur KSW (Other); Schweizer Lungenliga (Unknown)
Responsible Party: Principal Investigator, Anne-Kathrin Rausch, MSc, Zurich University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2015-0179
Record Dates: First submitted 2015-05-21; First posted 2015-05-27 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Usual Care (Active Comparator): outpatient pulmonary Rehabilitation program
  Interventions: Behavioral: Usual care
- Counseling (Experimental): outpatient pulmonary Rehabilitation program plus physical activity counseling
  Interventions: Behavioral: physical activity counseling

INTERVENTIONS:
Behavioral: physical activity counseling — 5 face-to-face sessions a 30 minutes during 12 weeks pulmonary rehabilitation program.
  Arms: Counseling
Behavioral: Usual care
  Arms: Usual Care

SUMMARY:
The purpose of this study is to investigate if a physical activity counseling program during pulmonary rehabilitation increases the physical activity level in daily life in patients with Chronic Obstructive Pulmonary Disease.

DETAILED DESCRIPTION:
Participants performed a 12 weeks outpatient pulmonary rehab (PR) according to guidelines. Participants allocated to intervention received PR plus physical activity (PA) counselling. PA counselling was performed using "motivational interviewing" techniques and was provided by two experiences physiotherapists independant to the rehab team. After PR and three months follow-up was evaluated if PA counselling during PR increases PA elvel (primary outcome: steps per day) in daily life.

Furthermore, individual, semi-structured interviews were performed in a subgroup of participants in order to gain more detailed information about barriers and enablers of participation in daily-life activities. Participants were invited to two interviews, one right after PR the other after 3 months follow up. A content analysis was performed.

ELIGIBILITY:
Inclusion Criteria:

* confirmed COPD (GOLD stages B-D) according to GOLD-guidelines

Exclusion Criteria:

* Mental or physical disability (mini-mental score <20) precluding informed consent or compliance with the protocol
* morphine medication
* Primary diagnosis of heart failure
* Uncontrolled arrhythmias causing symptoms or hemodynamic compromise
* Severe co-morbidity (acute coronary syndrome, unstable angina terminal renal failure, concomitant pulmonary embolism, very severe pneumonia: CURB65>3)
* Severe untreated arterial hypertension at rest (> 200 mm Hg systolic, > 120 mm Hg diastolic)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
number of steps per day | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hess, Dr med, Principal Investigator — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital, Winterthur, Switzerland

REFERENCES:
- [Derived] Rausch Osthoff AK, Beyer S, Gisi D, Rezek S, Schwank A, Meichtry A, Sievi NA, Hess T, Wirz M. Effect of counselling during pulmonary rehabilitation on self-determined motivation to be physically active for people with chronic obstructive pulmonary disease: a pragmatic RCT. BMC Pulm Med. 2021 Oct 12;21(1):317. doi: 10.1186/s12890-021-01685-2. PMID 34641819
- [Derived] Scheermesser M, Reicherzer L, Beyer S, Gisi D, Rezek S, Hess T, Wirz M, Rausch Osthoff AK. The Influence of Pulmonary Rehabilitation and Counselling on Perceptions of Physical Activity in Individuals with COPD - A Qualitative Study. Int J Chron Obstruct Pulmon Dis. 2021 Aug 14;16:2337-2350. doi: 10.2147/COPD.S315130. eCollection 2021. PMID 34421298
- [Derived] Rausch-Osthoff AK, Greco N, Schwank A, Beyer S, Gisi D, Scheermesser M, Meichtry A, Sievi N, Hess T, Wirz M. Effect of counselling during pulmonary rehabilitation on self-determined motivation towards physical activity in people with chronic obstructive pulmonary disease - protocol of a mixed methods study. BMC Pulm Med. 2017 Aug 17;17(1):115. doi: 10.1186/s12890-017-0457-8. PMID 28818057